CLINICAL TRIAL: NCT01549223
Title: A Randomized Controlled Trial of Standardized Versus Conventional Oxytocin and Uterotonic Agent Use for Cesarean Delivery
Brief Title: Oxytocin And Uterotonic Agent Use For Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Vice Chair, Faculty Development and Education; Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-P-002284
Record Dates: First submitted 2012-03-03; First posted 2012-03-09 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Uterine Atony; Hypotension
Keywords: Uterine Atony; Hypotension; Cesarean Delivery; Hemorrhage; Phenylephrine; Ephedrine
MeSH Terms: conditions — Uterine Inertia; Hypotension; Hemorrhage | interventions — Methylergonovine; carboprost tromethamine; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Care Group (Active Comparator): "Standard Care Group" (reflects current clinical regimen at BWH) will receive a 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request. The obstetrician and anesthesiologist will be asked to consider this infusion "oxytocin". If inadequate uterine tone exists in which the obstetrician desires alternative uterotonic agents, these will be provided on their request (e.g. methylergonovine maleate (methergine) 0.2 mg IM (intramuscular) or carboprost tromethamine (hemabate) 0.25 mg IM. The time of the requests will be recorded.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Interventions: Drug: Oxytocin Infusion
- Protocol Group (Active Comparator): "Protocol Group" will receive 3 mL syringes marked "study solution-oxytocin" which contain 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
  If inadequate uterine tone is noted at 9 min, the 1 mL syringe marked marked "study solution-9 min", containing methylergonovine maleate (methergine) 0.2mg, will be given IM.
  If inadequate uterine tone is noted at 12 min, the 1 mL syringe marked marked "study solution-12 min", containing carboprost tromethamine (hemabate) 0.25 mg, will be given IM.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Interventions: Drug: Oxytocin Bolus

INTERVENTIONS:
Drug: Oxytocin Infusion — 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request.
  Other Names: methylergonovine maleate (methergine) 0.2 mg IM; carboprost tromethamine (hemabate) 0.25 mg IM; misoprostol 600 mcg buccally
  Arms: Standard Care Group
Drug: Oxytocin Bolus — 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
  Other Names: methylergonovine maleate (methergine) 0.2 mg IM; carboprost tromethamine (hemabate) 0.25 mg IM; misoprostol 600 mcg buccally
  Arms: Protocol Group

SUMMARY:
The central objective of this study will be to evaluate a standardized, evidence-based regimen versus a conventional regimen for uterotonic drug dosing for elective cesarean delivery

The investigators primary hypothesis is that the proposed uterotonic drug regimen, when compared to conventional dosing regimen, during elective cesarean delivery will:

1. Reduce the overall amount of oxytocin and other uterotonic agents used to obtain satisfactory uterine tone.

Secondary outcomes to be evaluated will be:

1. Reduce the side effects associated with uterotonic drug use
2. Reduce the time to establishment and maintenance of adequate uterine tone

DETAILED DESCRIPTION:
The current guidelines for the administration of oxytocin during cesarean delivery are diverse, empiric, and vague. A stepwise, standardized, checklist driven algorithm for the use of oxytocin and other uterotonic agents during cesarean delivery is needed to guide practitioners in a clear and concise manner. This algorithm should encompass laboring and non-laboring women, as well as prophylactic and therapeutic uses of oxytocin and other uterotonic agents.

More specifically, the investigators believe that the following points should be incorporated into a protocol: 1) oxytocin should be used in initial doses of less than 5 IU; 2) oxytocin should not be administered as a rapid IV bolus; 3) an initial rapid infusion of oxytocin should be followed by a maintenance infusion; 4) higher initial and infusion doses of oxytocin offer no clinical benefit and should be avoided; and 5) if it appears that oxytocin is not producing effective uterine contractions, other uterotonic drugs acting via different pathways should be considered in a standardized way.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I or II health status
* Age between 18 and 50 yrs
* Singleton pregnancies in vertex position
* Elective (without prior labor) cesarean delivery with a planned lower uterine (pfannenstiel) incision

Exclusion Criteria:

* Conditions that predispose to uterine atony and postpartum hemorrhage

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Tsen, MD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care Group: "Standard Care Group" (reflects current clinical regimen at BWH) will receive a 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request. The obstetrician and anesthesiologist will be asked to consider this infusion "oxytocin". If inadequate uterine tone exists in which the obstetrician desires alternative uterotonic agents, these will be provided on their request (e.g. methylergonovine maleate (methergine) 0.2 mg IM (Intramuscular) or carboprost tromethamine (hemabate) 0.25 mg IM. The time of the requests will be recorded.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Oxytocin: 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request.
- Protocol Group: "Protocol Group" will receive 3 mL syringes marked "study solution-oxytocin" which contain 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
  If inadequate uterine tone is noted at 9 min, the 1 mL syringe marked marked "study solution-9 min", containing methylergonovine maleate (methergine) 0.2mg, will be given IM (Intramuscular).
  If inadequate uterine tone is noted at 12 min, the 1 mL syringe marked marked "study solution-12 min", containing carboprost tromethamine (hemabate) 0.25 mg, will be given IM.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Oxytocin: 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
Period: Overall Study
Arm/Group | Standard Care Group | Protocol Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Care Group: "Standard Care Group" (reflects current clinical regimen at BWH) will receive a 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request. The obstetrician and anesthesiologist will be asked to consider this infusion "oxytocin". If inadequate uterine tone exists in which the obstetrician desires alternative uterotonic agents, these will be provided on their request (e.g. methylergonovine maleate (methergine) 0.2 mg IM or carboprost tromethamine (hemabate) 0.25 mg IM. The time of the requests will be recorded.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Oxytocin: 500 mL bag of oxytocin (30 IU/500 mL) to be connected to the IV, and controlled per obstetrician request.
- Protocol Group: "Protocol Group" will receive 3 mL syringes marked "study solution-oxytocin" which contain 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
  If inadequate uterine tone is noted at 9 min, the 1 mL syringe marked marked "study solution-9 min", containing methylergonovine maleate (methergine) 0.2mg, will be given IM.
  If inadequate uterine tone is noted at 12 min, the 1 mL syringe marked marked "study solution-12 min", containing carboprost tromethamine (hemabate) 0.25 mg, will be given IM.
  If uterine tone remains inadequate at 15 min, misoprostol 600 mcg will be given buccally.
  Oxytocin: 3 IU oxytocin and be given IV at time of baby delivery (Time 0). Up to two additional syringes can be given at 3 and 6 mins until uterine tone adequate (as per obstetrician on graded scale).
- Total: Total of all reporting groups
Arm/Group | Standard Care Group | Protocol Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 40 years of age | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: 1. Amount of Oxytocin to Obtain Satisfactory Uterine Tone.
Description: Will measure total amount of oxytocin to achieve satisfactory uterine tone, as determined by the operating obstetrician.
Time Frame: Up to 15 min from time of infant delivery
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Standard Care Group | Protocol Group
Number analyzed (Participants) | 30 | 30
IU | 8.4 (4.8) | 4.0 (0.9)

2. Secondary Outcome: Side Effects (Hypotension, Flushing, Nausea and Emesis) Associated With Uterotonic Drug Use
Description: Number of subjects experiencing hypotension, flushing, nausea, and emesis reported after administration of uterotonic agents.
Time Frame: Up to 15 min from time of infant delivery
Population: All side effects: hypotension, flushing, nausea and emesis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Group | Protocol Group
Number analyzed (Participants) | 30 | 30
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Preoperatively until 6 hrs following cesarean delivery
Arm/Group | Standard Care Group | Protocol Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes